CLINICAL TRIAL: NCT03858998
Title: Reducing Post-Hospital Mortality in HIV-infected Adults in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1804019134; R01MH118107-01 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-03-01 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Management Intervention (Experimental): A 90-day case management intervention to link hospitalized HIV-infected participants with local HIV clinics.
  Interventions: Other: Case Management Intervention; Other: Control
- Control (Other): Current routine HIV care in Tanzania.
  Interventions: Other: Control

INTERVENTIONS:
Other: Case Management Intervention — A 90-day case management intervention to link hospitalized HIV-infected participants with local HIV clinics.
  Arms: Case Management Intervention
Other: Control — Current routine HIV care in Tanzania.

SUMMARY:
This research is being done to assess the efficacy of a case management intervention to improve the one year mortality rate of hospitalized, HIV-infected, Tanzanian adults.

DETAILED DESCRIPTION:
This research is being done to assess the efficacy of a case management intervention to improve the one year mortality rate of hospitalized, HIV-infected, Tanzanian adults. The study is being conducted at hospitals in Mwanza, Tanzania. 500 participants will be enrolled: 250 will be randomized to the case management intervention and 250 will randomized to routine clinical care. The case management intervention consists of 5 sessions over 90 days, and is designed to link hospitalized, HIV-infected patients to long term care at an HIV clinic. Participants will be followed for two years in order to evaluate primary and secondary study objectives.

Secondary outcome measures time frames have been updated to add the 24-month time point for consistency with the pre-specified endpoints in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* HIV-infected
* ART (anti-retroviral therapy) naïve or have been on ART but have not used ART for > 7 days
* Lives in the region of Mwanza
* Able to be referred to an HIV clinic inside the region of Mwanza
* Has mobile phone or access to mobile phone
* Planning to stay in the region of Mwanza for the next 24 months
* Able to speak Kiswahili or English
* Capable and willing to provide informed consent
* Willing to provide locator information and two designated contact persons
* Willing to have a home visits from a study team member

Exclusion Criteria

* Pregnant
* On anti-retrovirals at hospital admission and already linked to an HIV clinic
* Medical, psychiatric or psychological condition that, in the opinion of the site investigator, would interfere with completion of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Peck, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (16):
- Tanzania (16):
  - Busisi Health Center, Busisi, Mwanza Region
  - Magu District Hospital, Magu, Mwanza Region
  - Nyamilama Health Center, Nyamilama, Mwanza Region
  - Sengerema Health Center, Sengerema, Mwanza Region
  - Bugando Medical Center, Mwanza
  - Bukumbi Hospital, Mwanza
  - Buzuruga Health Center, Mwanza
  - Evangelical Lutheran Church in Tanzania (ELCT) Health Centre, Mwanza
  - Igoma Health Centre, Mwanza
  - Karume Health Centre, Mwanza
  - Kwimba District Hospital, Mwanza
  - Misungwi District Hospital, Mwanza
  - Nyamagana District Hospital, Mwanza
  - Sekou Toure Hospital, Mwanza
  - Sengerema District Hospital, Mwanza
  - Seventh Day Adventist (SDA) Health Centre, Mwanza

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include de-identified data on demographic characteristics, medical history, psychosocial measures, survival, HIV clinic linkage and retention, ART adherence, HIV viral loads, health economic variables and acceptability. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Therefore, we will make the dataset available to users under a data-sharing agreement that includes the following: a commitment to use the data for research purposes and not participant identification, commitment to securing the data with appropriate password protected IT practices, and a commitment to destroying the data after analyses are completed.
  For published data, the de-identified individual participant data that underlie the results reported in the article (text, tables, figured, appendices) will be available.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the protocol. Proposals should be directed to the Principal Investigator (rnp2002@med.cornell.edu).

REFERENCES:
- [Derived] Ayieko P, Willkens M, Issarow B, Deogratias D, Fitzgerald DW, Grosskurth H, Kisigo G, Okello E, Metsch LR, Peck RN, Kapiga S, Lee MH. Self-Efficacy and One-Year HIV Outcomes for Hospitalized People with HIV in Tanzania: A Mediation Analysis of the Daraja Clinical Trial. AIDS Behav. 2025 Nov 11:10.1007/s10461-025-04917-2. doi: 10.1007/s10461-025-04917-2. Online ahead of print. PMID 41214254
- [Derived] Okello ES, Peck RN, Issarow B, Kisigo G, Abel K, Malibwa D, Kabakama S, Charles M, Lee M, Rutachunzibwa T, Fitzgerald D, Ayieko P, Grosskurth H, Metsch LR, Kapiga S. "Ashamed of being seen in an HIV clinic": a qualitative analysis of barriers to engaging in HIV care from the perspectives of patients and healthcare workers in the Daraja clinical trial. BMC Public Health. 2025 Jan 7;25(1):69. doi: 10.1186/s12889-024-21231-z. PMID 39773172
- [Derived] Peck RN, Issarow B, Kisigo GA, Kabakama S, Okello E, Rutachunzibwa T, Willkens M, Deogratias D, Hashim R, Grosskurth H, Fitzgerald DW, Ayieko P, Lee MH, Murphy SM, Metsch LR, Kapiga S. Linkage Case Management and Posthospitalization Outcomes in People With HIV: The Daraja Randomized Clinical Trial. JAMA. 2024 Mar 26;331(12):1025-1034. doi: 10.1001/jama.2024.2177. PMID 38446792
- [Derived] Kisigo GA, Issarow B, Abel K, Hashim R, Okello ES, Ayieko P, Lee MH, Grosskurth H, Fitzgerald D, Peck RN, Kapiga S. A social worker intervention to reduce post-hospital mortality in HIV-infected adults in Tanzania (Daraja): Study protocol for a randomized controlled trial. Contemp Clin Trials. 2022 Feb;113:106680. doi: 10.1016/j.cct.2022.106680. Epub 2022 Jan 13. PMID 35032664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitalized people with HIV who were either not treated (antiretroviral-naïve) or had discontinued ART and were hospitalized for any reason were enrolled between March 2019 and February 2022.
Groups:
- Linkage Case Management Intervention: A 90-day case management intervention to link hospitalized HIV-infected participants with local HIV clinics.
- Enhanced Standard of Care: Current routine HIV care in Tanzania.
Period: Overall Study
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Started | 250 | 250
Completed | 250 | 250
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12) | 36 (11) | 37 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 194 | 384
  Male | 60 | 56 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 250 | 250 | 500
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 250 | 250 | 500
HIV/ART status [Count of Participants; unit: Participants]
  Newly diagnosed HIV | 211 | 191 | 402
  Previously diagnosed HIV and discontinued ART (≥ 7 days) | 39 | 59 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Deaths in the First 12 Months Post-hospitalization
Description: The number of participants who die in the first 12 months post-hospitalization will be recorded. Death will be determined by phone calls to relatives and will be confirmed by verbal autopsies, obituaries, hospital records, or death certificates.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
Participants | 43 | 42
Statistical Analysis 1: Comparison: Linkage Case Management Intervention vs Enhanced Standard of Care; Test type: Superiority; p = 0.91, Chi-squared; Risk Difference (RD) = 0.004, 95% CI 2-sided [-0.06 to 0.07] — Direction = Linkage minus SOC

2. Secondary Outcome: Number of Participants Who Attended HIV Clinic
Description: HIV clinic attendance will be monitored by review of HIV clinic records. HIV clinic attendance is defined as alive and attended clinic within a window of 90 days (+/- 45 days) around the time points.
Time Frame: 3, 6, 9,12, and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Case Management Intervention | Control
Number analyzed (Participants) | 250 | 250
Participants
  3 months | 215 | 187
  6 months | 190 | 160
  9 months | 180 | 158
  12 months | 180 | 158
  24 months | 161 | 143

3. Secondary Outcome: ART Adherence
Description: ART adherence will be assessed using the ACTG 4-Day ART Recall Questionnaire. Adherence will be calculated as a percentage, using 1 - (number of missed doses/number of prescribed doses).
Time Frame: 3, 6, 9, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percentage of ART adherence
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
percentage of ART adherence
  3 months | 95.1 (21.5) | 94.6 (22.0)
  6 months | 95.7 (19.5) | 91.6 (27.1)
  9 months | 90.9 (28.2) | 93.0 (25.0)
  12 months | 86.9 (33.3) | 77.8 (41.5)
  24 months | 85.0 (35.5) | 72.1 (44.7)

4. Secondary Outcome: Viral Suppression
Description: Suppressed viral load will be defined as a binary outcome based upon the WHO definition of viral suppression as a plasma HIV-1 RNA level <1000 copies/µl.
Time Frame: 12 and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
Participants
  12 months | 162 | 139
  24 months | 153 | 134

5. Secondary Outcome: Traditional Health Beliefs
Description: Traditional health beliefs will be assessed at baseline and after 12 months using the HIV Insights and Beliefs Scale, scored from 0 to 6, where higher scores indicate more traditional health beliefs. The minimum value is 0 and the maximum value is 6.
Time Frame: Baseline,12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
score on a scale
  Baseline | 0.53 (0.80) | 0.44 (0.79)
  12 months | 0.81 (0.80) | 0.89 (0.93)
  24 months | 1.10 (1.05) | 1.31 (1.34)

6. Secondary Outcome: Self-Efficacy
Description: Self-efficacy will be assessed at baseline and after 12 months using the HIV Adherence Self-Efficacy Scale, scored from 0 to 25, where higher scores indicate a higher level of self-efficacy.
Time Frame: Baseline, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
score on a scale
  Baseline | 22.42 (2.72) | 22.39 (2.86)
  12 months | 22.65 (3.68) | 21.47 (5.39)
  24 months | 22.48 (4.96) | 20.50 (6.64)

7. Secondary Outcome: Stigma
Description: Stigma will be assessed at baseline and after 12 months using questions based off the AIDS-Related Stigma Scale, scored from 0 to 8, where higher scores indicate a higher level of perceived stigma.
Time Frame: Baseline, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
score on a scale
  Baseline | 2.32 (0.92) | 2.28 (0.91)
  12 months | 2.12 (0.87) | 2.24 (0.88)
  24 months | 2.16 (0.94) | 2.27 (0.92)

8. Secondary Outcome: Social Support
Description: Social support will be assessed at baseline and after 12 months using the SPS-10 Scale, scored from 0 to 40, where higher scores indicate a higher level of social support.
Time Frame: Baseline, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
score on a scale
  Baseline | 34.84 (4.66) | 34.74 (4.35)
  12 months | 33.02 (5.14) | 32.59 (4.60)
  24 months | 33.16 (4.74) | 31.66 (5.78)

9. Secondary Outcome: Perceived Need for HIV Services
Description: Perceived need for HIV services will be assessed at baseline and after 12 months using the ART Medications Attitude Scale, scored from 0 to 4, where higher scores indicate a lower perceived need for HIV services.
Time Frame: Baseline, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
score on a scale
  Baseline | 1.90 (0.30) | 1.94 (0.30)
  12 months | 1.85 (0.37) | 1.86 (0.41)
  24 months | 1.90 (0.31) | 1.91 (0.36)

10. Secondary Outcome: SF-12 Health Survey: Physical and Mental Health
Description: Physical weakness will be assessed at baseline and after 12 months using the SF-12 Health Survey. The SF-12 measures physical health (physical component score (PCS)), scored from 0 to 100, and mental health (mental component score (MCS)), scored from 0 to 100, with higher scores indicating greater physical and mental health.
Time Frame: Baseline, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
score on a scale
  Physical component score (PCS )- Baseline | 37.52 (9.13) | 37.15 (9.04)
  Mental component score (MCS) - Baseline | 45.08 (11.87) | 44.76 (11.92)
  PCS - 12 months | 50.59 (8.31) | 51.15 (8.06)
  MCS - 12 months | 49.64 (12.79) | 50.42 (11.85)
  PCS - 24 months | 50.91 (8.23) | 50.92 (7.59)
  MCS - 24 months | 51.13 (12.98) | 51.29 (11.85)

11. Secondary Outcome: Acceptability
Description: Qualitative interviews will be conducted with a sub-set of participants to evaluate the acceptability of the intervention. The acceptability of the Daraja intervention was defined as a binary outcome based on the results of the qualitative interviews. The sub-set will be comprised of 20 intervention participants, 20 routine care control participants, and 20 health care workers (nurses and physicians). Health care workers were not enrolled as participants in the trial nor randomized to a study arm.
Time Frame: 12 and 24 months
Population: We assessed the acceptability of the Daraja intervention across the study groups through qualitative interviews. The subset of participants for qualitative interviews were purposively selected from the list of participants who had completed 12 months from enrollment. We selected 20 intervention participants, 20 control participants and 20 healthcare workers providing care to people with HIV. Health care workers were not enrolled as participants in the trial nor randomized to a study arm.
Measure: Count of Participants; unit: Participants
Groups:
- Health Care Workers: Health care workers involved with care of hospitalized people with HIV.
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care | Health Care Workers
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Acceptability -12 months | 20 | 20 | 20
  Acceptability - 24 months | 20 | 20 | 20

12. Secondary Outcome: Incremental Cost of the Intervention
Description: A microcosting analysis was conducted to identify the resources needed to implement and sustain the Daraja intervention and estimate the associated costs. Resource identification was accomplished primarily through in-person site visits and semi-structured interviews with relevant personnel. Nationally representative unit costs were assigned to the relevant resources. Resources were categorized as fixed start-up, time-dependent, or variable, and contextualized as being required for implementation or sustainment. The intervention implementation period was defined as the first 12 months following start-up, and consisted of the resources in all 3 of the aforementioned categories, and the sustainment period is intended to reflect a typical year following the implementation period, and consists of time-dependent and variable resources, given that the costs associated with fixed start-up resources become negligible over time. Incremental cost was reported as a number in 2023 USD.
Time Frame: 12 months
Measure: Number; unit: US dollar
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 250 | 250
US dollar
  Year 1 costs, per client | 22 | 0
  Annual sustainment costs, per client | 17 | 0

13. Secondary Outcome: Cost Per Life Saved
Description: The difference in costs between the arms from the healthcare perspective will be compared to the observed difference in survival between the arms to calculate incremental cost per life saved. Parametric methods based on parameters obtained from bootstrapping will be used to estimate an acceptability curves, which will illustrate the probability that the intervention is a good value for different willingness-to-pay thresholds
Time Frame: 12 months
Population: This measure could not be calculated because it assumed an outcome that was not observed.
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: All-cause mortality was the primary outcome of this trial.
Arm/Group | Linkage Case Management Intervention | Enhanced Standard of Care
All-Cause Mortality (participants affected / at risk) | 43/250 | 42/250
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/250
Other Adverse Events (participants affected / at risk) | 0/250 | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT03858998/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT03858998/SAP_001.pdf